CLINICAL TRIAL: NCT02712541
Title: Caregiver Burden and Wellbeing in Relatives of Intensive Care Unit Patients
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Stockholm South General Hospital (Other); Uppsala University Hospital (Other); Region Örebro County (Other)
Responsible Party: Principal Investigator, Peter Sackey, Senior Consultant, Associate Professor, Karolinska University Hospital
Other Study IDs: EPN Dnr 2015/1799-31 (b)
Record Dates: First submitted 2016-02-05; First posted 2016-03-18 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Social Responsibility
Keywords: Caregiver burden Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether there is an association between adverse physical and/or psychological outcome in ICU survivors and the caregiver burden for their relatives.

We hypothesize that relatives to ICU survivors with an incomplete physical and/or psychological recovery three months after ICU stay report a higher caregiver burden.

DETAILED DESCRIPTION:
This is a sub-study to the multicenter "PROGRESS study". Details of the PROGRESS study have been described elsewhere. Briefly, an observational study including 600-1000 adult ICU patients from ten European hospitals will be followed up during three months to identify potential risk factors for physical and psychological problems.

The sub-study is conducted in four Swedish hospitals (Karolinska University Hospital Solna, Södersjukhuset, Stockholm, Örebro University Hospital and Akademiska University Hospital in Uppsala). Relatives to patients included in the PROGRESS study, who give informed consent to participate are consecutively included in the study.

Consenting participants (relatives) will be approached after inclusion of the patient and asked to estimate their own health related quality of life (HRQOL) 2 weeks prior to the time point for patient ICU admission through a HRQOL questionnaire. This self-reported HRQOL data will be used as proxy for baseline data. Three months after ICU discharge, relatives to ICU survivors will receive the following questionnaires by postal mail; Caregiver Burden Index, HRQOL questionnaire, a questionnaire screening for symptoms of anxiety and depression and a questionnaire screening for symptoms of posttraumatic stress.

The relatives will also be asked to state the number of working days lost due to caretaking of the ICU survivor.

ICU survivors' physical and psychological outcome, assessed with BI, SF-36, PTSS-14 and HADS three months after ICU discharge, obtained in the main PROGRESS study, will be compared with relatives' reported caregiver burden.

Secondary outcomes are associations between caregiver burden and reported health-related quality of life between baseline and 3 months after ICU discharge, frequency of symptoms of anxiety, depression and posttraumatic stress 3 months post ICU discharge and number of working days lost because of their relative's critical illness.

ELIGIBILITY:
Inclusion Criteria:

1. Relatives are considered eligible if they are a) partner to the patient b) adult children, siblings, parents or close friend that share household with the ICU survivor

Exclusion Criteria:

1. Non-Swedish-speaking
2. Overt or documented cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Relative living together with a patient included in the study PROGRESS-ICU.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Caregiver burden Index score | Three months after patients' discharge from the ICU
  Score compared between nearest of kin to patients with good or poor physical or psychological outcome (obtained in the main PROGRESS-ICU Study), three months after ICU discharge

SECONDARY OUTCOMES:
Short Form-36 | Three months after patients' ICU discharge
  Relation between Caregiver burden Index scores and mental component score in SF-36
Hospital Anxiety and Depression Scale | Three months post ICU discharge
  Relation between outcomes in patients and scores in nearest of kin
Posttraumatic stress symptoms Inventory - 14 | Three months post ICU discharge
  Relation between patients outcome and nearest of kin scores

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sackey, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (4):
- Sweden (4):
  - Örebro Universitetssjukhus, Örebro
  - Dept of Anesthesiology, Surgical Services and Intensive Care Medicine, Karolinska University Hospital, Stockholm
  - Stockholm South Hospital, Stockholm
  - Dept of Anesthesia and Intensive Care, Uppsala Akademiska, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided